CLINICAL TRIAL: NCT05508373
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Recombinant Fully Human Anti-CD39 Monoclonal Antibody JS019 in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability,JS019 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Kebo Ruijun Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS019-002-I
Record Dates: First submitted 2022-08-10; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: dose level：0.3mg/kg (Experimental): Dose Escalation: 0.3mg/kg, IV infusion, every 3 weeks (q3w).
  Interventions: Biological: JS019
- Dose Escalation: dose level：1 mg/kg (Experimental): Dose Escalation: 1 mg/kg IV infusion, every 3 weeks (q3w).
  Interventions: Biological: JS019
- Dose Escalation: dose level：3 mg/kg (Experimental): Dose Escalation: 3 mg/kg IV infusion, every 3 weeks (q3w).
  Interventions: Biological: JS019
- Dose Escalation: dose level：10 mg/kg (Experimental): Dose Escalation: 10 mg/kg IV infusion, every 3 weeks (q3w).
  Interventions: Biological: JS019

INTERVENTIONS:
Biological: JS019 — Four dose levels are preset: 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg. The subjects are treated with JS019 by intravenous infusion, once every 3 weeks (Q3W). A treatment cycle is 21 days, and the DLT observation period is 21 days after the first administration.

SUMMARY:
This is a phase 1 clinical study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of JS019 as monotherapy in patients with advanced malignant solid tumors The study includes JS019 monotherapy dose escalation, dose expansion stages to investigate the safety, tolerability, pharmacokinetics and preliminary anti-tumor efficacy of JS019 as monotherapy.

DETAILED DESCRIPTION:
Monotherapy Dose Escalation Stage:

In this stage, the safety and tolerability, PK characteristics, immunogenicity and pharmacodynamics characteristics of JS019 are investigated. Four dosage groups are preset: 0.3 mg/kg, 1 mg/kg, 3 mg/kg and 10 mg/kg. The drug is administered intravenously every 3 weeks (Q3W). A treatment cycle is 21 days, with a DLT observation period of 21 days after the initial administration. The incremental dose and dosing interval may be adjusted as necessary during the study based on safety, PK, and other results obtained

Monotherapy Dose Expansion Stage:

According to RP2D of JS019 single drug dose, 3-5 specific tumor types are selected for indication expansion, and about 8-12 patients are enrolled for each indication. Tumor types and additional cases could be selected according to the specific situation in the trial process. It is planned to expand the cohort of lung cancer, pancreatic cancer, sarcoma, hepatocellular carcinoma, cholangiocarcinoma and other solid tumors to explore the efficacy and safety of JS019 single drug. The specific cohort will be adjusted according to the results of previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and willing to sign the Informed Consent Form;
2. Male or female aged 18~75 years (included);
3. Patients with pathologically confirmed advanced malignant solid tumors
4. Failed or unsuitable for standard treatment;
5. Eastern Cooperative Oncology Group (ECOG) physical fitness score: 0~1;
6. Expected survival period ≥ 12 weeks;
7. At least one measurable lesion according to criteria RECIST v1.1 ;

Exclusion Criteria:

1. Patients with known hypersensitivity to the components of JS019;
2. Patients who have received the treatment with anti-CD39 antibodies or inhibitors;
3. Patients who participated in other clinical studies within 4 weeks prior to the first administration of JS019, except patients are in the follow-up period of observational (non-interventional) clinical study or interventional study;
4. Patients who have received major surgery within 4 weeks before the first dose or expected to undergo major surgery during the study (as judged by the investigator) or are in the recovery period from surgery;
5. Patients who have received anti-tumor therapy, such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, or biological therapy, within 4 weeks or 5 half-lives of the therapy (whichever is shorter) prior to the first dose of JS019. Patients who have received traditional Chinese medicine or Chinese patent medicine preparations with anti-tumor indications within 2 weeks before the first dose of JS019. Can accept hormone therapy for non-tumor-related diseases (such as insulin therapy for diabetes and hormone replacement therapy, etc.);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Safety Incidence of DLT severity of adverse events (AEs) and serious adverse events (SAEs)and tolerability | 2 years
  Incidence of DLT, incidence and severity of adverse events (AE) and severe adverse events (SAE), clinically significant abnormal laboratory changes and other tests
Maximum Tolerated Dose (MTD) or Optimal Biological Effect Dose (OBD) and Phase II study recommended dose (RP2D) | 2 years
  The safety, pharmacokinetic and preliminary efficacy data of the comprehensive dose escalation were determined. When MTD/OBD is determined, MTD/OBD is usually used as RP2D.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | 2 years
  Drug concentrations in individual subjects at different time points after administration
Immunogenicity | 2 years
  Incidence of anti-drug antibodies (ADA), titer of ADA-positive samples.
Pharmacodynamics （PD） | 2 years
  CD39 receptor occupancy in peripheral blood.
Objective response rate (ORR) | 2 years
  The percentage of cases with remission (PR + CR) after treatment was assessable
Duration of response (DOR) | 2 years
  The time from the first assessment of CR or PR to the first assessment of PD or death due to any cause.
Disease control rate (DCR) | 2 years
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
Time to response (TTR) | 2 years
  time from the start of treatment to progression of diease.
Progression-free survival (PFS) | 2 years
  PFS is defined as time from the start of treatment to progression of disease or death.
Overall survival (OS) | 2 years
  Overall survival is defined as time from the start of treatment until death due to any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided